CLINICAL TRIAL: NCT01275781
Title: A Phase 1, Open-Label, Non-randomized, Single-Center Study to Assess Distribution, Metabolism and Excretion After [14C]-Labelled Intravenous Administration of AZD9742 as a 2-hour Infusion to Healthy Male Volunteers
Brief Title: Study in Healthy Males to Assess Distribution, Metabolism, and Excretion of Radio-labelled AZD9742 Administered as a 2-hour Infusion
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to the local Radiation Safety Committee refusing to approve it.
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Medical Director, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D2690C00009
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Phase 1; healthy male volunteers; radioactivity; excretion; metabolism; AZD9742; amount of radioactive AZD9742 in urine, feces, and vomitus (if appropriate)
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): [14C]-AZD9742 1000 mg intravenous over 2 hours
  Interventions: Drug: [14C]-AZD9742

INTERVENTIONS:
Drug: [14C]-AZD9742 — 1000 mg intravenous over 2 hours

SUMMARY:
The purpose of this study is to assess distribution, metabolism, and excretion of radio-labelled AZD9742 administered as a 2-hour infusion to healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers age 55 years or older on Day 1, body weight >50 kg, body mass index (BMI) between 18 kg/m2 and 30 kg/m2
* Regular bowel movements, at least once per day (self reported)
* Volunteers must be willing to have intravenous (IV) and blood sampling from either arm.
* Volunteers should ensure that their partners of child-bearing potential use a reliable method of contraception, as well as using a barrier method themselves.

Exclusion Criteria:

* History of any clinically significant disease or abnormalities, including history or presence of gastrointestinal, hepatic, renal disease or any other condition known to interfere with metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product
* Current smokers or those who have smoked or used nicotine products within the previous 30 days
* History of alcohol abuse or excessive intake of alcohol
* Participation in more than 1 other radiolabeled investigational study drug trial within 1 year prior to check-in. The previous radiolabeled study drug had to be received more than 6 months prior to check-in and the total exposure from this study and the previous study must be within the CFR recommended levels considered safe (per 21 CRF 362.1, less than 5,000 mrem whole body annual exposure).

Min Age: 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
To characterize the distribution and elimination of AZD9742 and total 14C radioactivity in healthy volunteers following a single 1000 mg intravenous (IV) dose of [14C]-AZD9742 administered as a 2-hour infusion. | Range of 12 hours pre dose to 168 hours post dose
  12 hours pre dose to 168 hours post dose of the treatment period if the patient meets discharge criteria. If the patient does not meet discharge criteria after 168 hours post dose, additional 24 hour collections up to 7 additional days or until discharge criteria are met, whichever occurs first.
To evaluate the excretion of 14C (mass balance) in urine and feces after a single 1000 mg intravenous (IV) dose of [14C]-AZD9742 administered as a 2-hour infusion. | Range of 12 hours pre dose to 168 hours post dose
  12 hours pre dose to 168 hours post dose of the treatment period if the patient meets discharge criteria. If the patient does not meet discharge criteria after 168 hours post dose, additional 24 hour collections up to 7 additional days or until discharge criteria are met, whichever occurs first.

SECONDARY OUTCOMES:
Safety of AZD9742 after a single intravenous 14C administration of AZD9742, by assessing a panel of measures: Adverse Events, vital sign evaluations, physical examination, electrocardiograms (ECG) and clinical laboratory parameters.
To explore and establish the metabolite profiles in plasma and excreta; where possible the identity of metabolites will be determined. | Immediately prior to the end of the infusion, 4 hours after the end of the infusion and 24 hours after the start of the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — AstraZeneca; Ralph Schutz, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States